CLINICAL TRIAL: NCT00677313
Title: An Open-Label Treatment Protocol to Provide Metreleptin for the Treatment of Diabetes Mellitus and/or Hypertriglyceridemia Associated With Lipodystrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MB002-002; FHA101 (Other: Amylin)
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-02

CONDITIONS: Lipodystrophy
Keywords: metreleptin; leptin; Amylin; diabetes mellitus; hypertriglyceridemia; lipodystrophy
MeSH Terms: conditions — Lipodystrophy; Diabetes Mellitus; Hypertriglyceridemia | interventions — metreleptin

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: metreleptin

INTERVENTIONS:
Drug: metreleptin — metreleptin injection

SUMMARY:
This is an open-label study to provide metreleptin for the treatment of diabetes mellitus and/or hypertriglyceridemia associated with lipodystrophy. This study intends to provide guidance to investigators with respect to identification of appropriate subjects for metreleptin treatment, guidance on metreleptin dosing, and collection of safety and efficacy data following metreleptin treatment in this population

ELIGIBILITY:
Inclusion Criteria:

* Is male or female ≥5 years old
* If female of childbearing potential (including perimenopausal women who have had a menstrual period within one year):

  1. Not breastfeeding
  2. Negative pregnancy test result
  3. Must practice and be willing to continue to practice appropriate birth control (defined as a method which results in a low failure rate, i.e., less than 1% per year, when used consistently and correctly, such as implants, injectables, oral contraceptives, some intrauterine contraceptive devices, sexual abstinence, tubal ligation, or a vasectomized partner) during the entire duration of the study (Double barrier methods including the use of female diaphragm and male condom with spermicide can also be used.)
* Has physician-confirmed lipodystrophy as defined by evidence of generalized (whole body) or partial (limbs) loss of body fat outside the range of normal variation
* Has been diagnosed with at least one of the following 2 metabolic disorders:

  1. Diabetes Mellitus
  2. Hypertriglyceridemia as defined by fasting triglyceride concentrations >200 mg/dL
* If ≥18 years of age, is able to read, understand, and sign the Informed Consent Form (ICF) and an Authorization to Use and Disclose Protected Health Information form, communicate with the investigator, and understand and comply with protocol requirements
* If <18 years of age, has a parent or legal guardian to read and understand the ICF and Child Assent Form, communicate with the investigator, and understand and comply with protocol requirements. Adolescent subjects must also read and understand the Child Assent Form; if the child is too young or unable to read, then the Child Assent Form must be explained to the child.

Exclusion Criteria:

* Has been diagnosed with HIV infection
* Has known infectious liver disease
* Has known allergies to E. coli-derived proteins or hypersensitivity to any component of study treatment

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
To provide metreleptin, an investigational medication, under a treatment protocol to subjects with lipodystrophy that is associated with diabetes mellitus and/or hypertriglyceridemia | open ended

SECONDARY OUTCOMES:
To monitor the safety and tolerability of metreleptin in subjects with lipodystrophy that is associated with diabetes mellitus and/or hypertriglyceridemia | open ended
Information on the efficacy of metreleptin as assessed by its effects on fasting triglyceride concentrations, HbA1c, and fasting glucose concentrations in subjects with lipodystrophy that is associated with diabetes mellitus and/or hypertriglyceridemia | open ended

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- United States (5):
  - Research Site, Santa Barbara, California
  - Research Site, Chicago, Illinois
  - Research Site, Ann Arbor, Michigan
  - Local Institution, Reno, Nevada
  - Research Site, Greenville, North Carolina

REFERENCES:
- [Derived] Meral R, Malandrino N, Walter M, Neidert AH, Muniyappa R, Oral EA, Brown RJ. Endogenous Leptin Concentrations Poorly Predict Metreleptin Response in Patients With Partial Lipodystrophy. J Clin Endocrinol Metab. 2022 Mar 24;107(4):e1739-e1751. doi: 10.1210/clinem/dgab760. PMID 34677608
- [Derived] Ajluni N, Dar M, Xu J, Neidert AH, Oral EA. Efficacy and Safety of Metreleptin in Patients with Partial Lipodystrophy: Lessons from an Expanded Access Program. J Diabetes Metab. 2016 Mar;7(3):659. doi: 10.4172/2155-6156.1000659. Epub 2016 Mar 23. PMID 27642538
- [Derived] Chan JL, Koda J, Heilig JS, Cochran EK, Gorden P, Oral EA, Brown RJ. Immunogenicity associated with metreleptin treatment in patients with obesity or lipodystrophy. Clin Endocrinol (Oxf). 2016 Jul;85(1):137-49. doi: 10.1111/cen.12980. Epub 2016 Feb 2. PMID 26589105
- [Derived] Safar Zadeh E, Lungu AO, Cochran EK, Brown RJ, Ghany MG, Heller T, Kleiner DE, Gorden P. The liver diseases of lipodystrophy: the long-term effect of leptin treatment. J Hepatol. 2013 Jul;59(1):131-7. doi: 10.1016/j.jhep.2013.02.007. Epub 2013 Feb 21. PMID 23439261
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx